CLINICAL TRIAL: NCT05868187
Title: CanRestoreFunction: Cancer-Related Fatigue Management
Brief Title: CanRestoreFunction Cancer-related Fatigue ( CRF )
Acronym: CRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: University of Dayton (Other)
Responsible Party: Principal Investigator, Anne Fleischer, Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRP - 503
Record Dates: First submitted 2023-02-07; First posted 2023-05-22 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Breast Neoplasm
Keywords: cancer-related fatigue; breast cancer; exercise; problem-solving; online interactive education
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise, Problem-Solving and Education (Experimental): Individualized exercise program Weekly Goals setting and problem-solving session to create a weekly action plan Four Assigned interactive educational modules
  Interventions: Behavioral: Exercise, Problem-Solving Session and Education
- Usual Care (No Intervention): Participants will complete their daily routines as they typically do.

INTERVENTIONS:
Behavioral: Exercise, Problem-Solving Session and Education — Complete assigned exercises three times a week Complete Action plan co-developed Complete part or all of one of the four interactive educational modules
  Arms: Exercise, Problem-Solving and Education

SUMMARY:
The goal of this randomized control trial is to determine if participating in an 8-week online cancer-related fatigue management intervention consisting of individualized exercise program, one-on-one goal setting and action plan development and interactive educational module will significantly reduce the perception of cancer-related fatigue, improve the quality of life, improve perceived cognition, and perceived function of breast cancer compared to a wait-list control group. The aim the project is to determine if an online cancerrelated fatigue management program is associated with 1. A decrease in cancer-related fatigue. 2. An improved perception of their ability and satisfaction in completing important activities 3. Greater quality of life. 4. Improved mobility 5. Improved perceived cognition

ELIGIBILITY:
Inclusion Criteria:

* been diagnosed with any type of cancer within 5 years of enrollment,
* received chemotherapy and/or radiation therapy
* have access to mobile device or computer
* have basic computer or mobile device skills,
* have a significant level of fatigue defined as >3 on 0-10 scale using the Oneitem Fatigue Scale

Exclusion Criteria:

* have metastatic cancer (Stage 4),
* do not have a signed medical release by their physician or physician extender indicating that the participant can safely participate in the exercise program,
* chronic fatigue prior to cancer diagnosis, such as fibromyalgia
* are unable to follow verbal or written assessment instructions, are non-English speaking

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Brief Fatigue Inventory | Baseline
  This 9-item scale assesses the severity and interference of fatigue based on a 0 (no fatigue) to 10 (greatest fatigue) scale
Brief Fatigue Inventory | 4-week
  This 9-item scale assesses the severity and interference of fatigue based on a 0 (no fatigue) to 10 (greatest fatigue) scale
Brief Fatigue Inventory | 8-week
  This 9-item scale assesses the severity and interference of fatigue based on a 0 (no fatigue) to 10 (greatest fatigue) scale

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure | Baseline
  The OT administers the COPM, which is a semi-structured interview to understand the routine activities that the participant completes daily, specifically their self-care, leisure, and social activities. The participant rates the importance of each of the activities using a 0 to 10 scale. Zero indicates "no importance" and 10 indicates "very important." Then the participant separately rates their perception of how well they currently perform each of the important activities and how satisfied they are with their performance using a 0 to 10 scale. Zero indicates that "they are not able to perform" or "they are not satisfied" and 10 indicates that "they are able to perform the activity well" or "they are very satisfied."
Canadian Occupational Performance Measure | 4-week
  The OT administers the COPM, which is a semi-structured interview to understand the routine activities that the participant completes daily, specifically their self-care, leisure, and social activities. The participant rates the importance of each of the activities using a 0 to 10 scale. Zero indicates "no importance" and 10 indicates "very important." Then the participant separately rates their perception of how well they currently perform each of the important activities and how satisfied they are with their performance using a 0 to 10 scale. Zero indicates that "they are not able to perform" or "they are not satisfied" and 10 indicates that "they are able to perform the activity well" or "they are very satisfied."
Canadian Occupational Performance Measure | 8-week
  The OT administers the COPM, which is a semi-structured interview to understand the routine activities that the participant completes daily, specifically their self-care, leisure, and social activities. The participant rates the importance of each of the activities using a 0 to 10 scale. Zero indicates "no importance" and 10 indicates "very important." Then the participant separately rates their perception of how well they currently perform each of the important activities and how satisfied they are with their performance using a 0 to 10 scale. Zero indicates that "they are not able to perform" or "they are not satisfied" and 10 indicates that "they are able to perform the activity well" or "they are very satisfied."
Functional Assessment of Chronic Illness Therapy-Fatigue | Baseline
  This 40-item 5-point Likert scale (0=Not at all 1=A little bit 2=Somewhat 3= Quite a bit 4=Very much) evaluates quality of life in individuals with fatigue as measured in 5 domains: physical, social/family, emotional, functional well-being, and fatigue. Higher scores reflect greater quality of life
Functional Assessment of Chronic Illness Therapy-Fatigue | 4-weeks
  This 40-item 5-point Likert scale (0=Not at all 1=A little bit 2=Somewhat 3= Quite a bit 4=Very much) evaluates quality of life in individuals with fatigue as measured in 5 domains: physical, social/family, emotional, functional well-being, and fatigue. Higher scores reflect greater quality of life
Functional Assessment of Chronic Illness Therapy-Fatigue | 8-weeks
  This 40-item 5-point Likert scale (0=Not at all 1=A little bit 2=Somewhat 3= Quite a bit 4=Very much) evaluates quality of life in individuals with fatigue as measured in 5 domains: physical, social/family, emotional, functional well-being, and fatigue. Higher scores reflect greater quality of life
PROMIS Cognitive Function Ability 8a | Baseline
  This 8-item 5-point Likert scale [Never, Rarely (Once) Sometimes (Two or three times) Often (About once a day) Very often (Several times a day)] evaluates patient-perceived cognitive abilities, its interference with daily functioning, whether other people observe cognitive impairments, and its impact on quality of life
PROMIS Cognitive Function Ability 8a | 4-weeks
  This 8-item 5-point Likert scale [Never, Rarely (Once) Sometimes (Two or three times) Often (About once a day) Very often (Several times a day)] evaluates patient-perceived cognitive abilities, its interference with daily functioning, whether other people observe cognitive impairments, and its impact on quality of life
PROMIS Cognitive Function Ability 8a | 8-weeks
  This 8-item 5-point Likert scale [Never, Rarely (Once) Sometimes (Two or three times) Often (About once a day) Very often (Several times a day)] evaluates patient-perceived cognitive abilities, its interference with daily functioning, whether other people observe cognitive impairments, and its impact on quality of life
Promis Applied Cognitive Abilities 8a | Baseline
  This 8-item 5-point Likert scale [Not at all A little bit, Somewhat, Quite a bit, Very much] evaluates the patient-perceived cognitive deficits
Promis Applied Cognitive Abilities 8a | 4-weeks
  This 8-item 5-point Likert scale [Not at all A little bit, Somewhat, Quite a bit, Very much] evaluates the patient-perceived cognitive deficits
Promis Applied Cognitive Abilities 8a | 8-weeks
  This 8-item 5-point Likert scale [Not at all A little bit, Somewhat, Quite a bit, Very much] evaluates the patient-perceived cognitive deficits
6-minute walk test | Baseline
  Participants completes a 6-minute walk at their chosen pace and with permitted standing rest breaks
6-minute walk test | 4-weeks
  Participants completes a 6-minute walk at their chosen pace and with permitted standing rest breaks
6-minute walk test | 8-weeks
  Participants completes a 6-minute walk at their chosen pace and with permitted standing rest breaks
30 second sit to stand | Baseline
  Participants are seated in a standard height fixed chair without armrests, which is placed against a wall. They will move from sitting to standing and back to sitting position, with arms crossed against chest. The number of complete stands and sits
30 second sit to stand | 4-weeks
  Participants are seated in a standard height fixed chair without armrests, which is placed against a wall. They will move from sitting to standing and back to sitting position, with arms crossed against chest. The number of complete stands and sits
30 second sit to stand | 8-weeks
  Participants are seated in a standard height fixed chair without armrests, which is placed against a wall. They will move from sitting to standing and back to sitting position, with arms crossed against chest. The number of complete stands and sits
Average number of steps | Week 1
  Fitbit will track the number of steps that the participants takes each day
Average number of steps | Week 2
  Fitbit will track the number of steps that the participants takes each day
Average number of steps | Week 3
  Fitbit will track the number of steps that the participants takes each day
Average number of steps | Week 4
  Fitbit will track the number of steps that the participants takes each day
Average number of steps | Week 5
  Fitbit will track the number of steps that the participants takes each day
Average number of steps | Week 6
  Fitbit will track the number of steps that the participants takes each day
Average number of steps | Week 7
  Fitbit will track the number of steps that the participants takes each day
Average number of steps | Week 8
  Fitbit will track the number of steps that the participants takes each day
Average heart rate | Week 1
  Fitbit will track daily heart rate of each participant
Average heart rate | Week 2
  Fitbit will track daily heart rate of each participant
Average heart rate | Week 3
  Fitbit will track daily heart rate of each participant
Average heart rate | Week 4
  Fitbit will track daily heart rate of each participant
Average heart rate | Week 5
  Fitbit will track daily heart rate of each participant
Average heart rate | Week 6
  Fitbit will track daily heart rate of each participant
Average heart rate | Week 7
  Fitbit will track daily heart rate of each participant
Average heart rate | Week 8
  Fitbit will track daily heart rate of each participant

CONTACTS AND LOCATIONS:
Overall Officials: Anne Fleischer, Ph.D, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States